CLINICAL TRIAL: NCT04668430
Title: Imaging for the Generation of Personalized Biomechanical Models of the Musculoskeletal System Before and After Surgery
Brief Title: Evaluation of Personalized Biomechanical Models of the Musculoskeletal System Before and After Orthopedic Surgeries
Acronym: OrthosimPro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02124-53
Record Dates: First submitted 2020-11-12; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-04

CONDITIONS: Orthopedic Disorder
Keywords: computer simulation; orthopedic surgical procedures; Multimodal Imaging; gait analysis
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Other): Patients for whom orthopedic surgery is indicated and planned among :
  * Tibial valgus osteotomy
  * Supra-malleolar osteotomy
  * Hallux osteotomy for hallux valgus
  * Total knee arthroplasty
  * Total ankle arthroplasty
  * Ankle arthrodesis
  * Hallux arthrodesis
  * Rear foot torque arthrodesis
  * Inverted shoulder prosthesis
  * Anterior lumbar interbody arthrodesis
  Interventions: Other: imaging and motion analysis

INTERVENTIONS:
Other: imaging and motion analysis — performing a set of imaging and motion analysis tests before and after orthopedic surgery without modifying the operative indication or the pre- and post-operative management.

SUMMARY:
Advances in biomechanical modeling of musculoskeletal systems make it possible to consider the use of a digital clone of a patient to test surgical procedure before carrying it out on the patient himself.

The study aims at evaluating the design and simulation procedure of anatomical and functional pre and post surgical patient-specific numerical models.

DETAILED DESCRIPTION:
The general research framework is focused on predicting the functional outcome of orthopaedic surgery for a given patient.

Since surgery is an invasive and irreversible procedure, it may be useful to carry out surgical simulations on a digital clone before performing them on the real patient.

This simulation would therefore be a tool for optimized surgical planning, based on a realistic functional objective.

The investigators' work in the design and evaluation of biomechanical models is now applicable to orthopedic surgery.

So, it is necessary to verify that the digital procedures allowing the realization of virtual surgical gestures are comparable to the procedures actually applied to the patient.

Thus, a first retrospective study (Imaging for the generation of personalized biomechanical models of the musculoskeletal system before and after surgery - ORTHOSIM Retrospective) Clinical Trial N° NCT03835000, is in progress in order to validate the possibility of creating pre- and post-operative anatomical digital clones. The aim of this prospective study is to integrate the functional characteristics of the patient before and after surgery with the objective of dynamic validation of the biomechanical models created.

OrthosimPro is a bi-centric, longitudinal and prospective study.

10 patients needing orthopedic surgery will be enrolled after being informed about the study and potential risks. They will give written informed consent.

This study will not modify :

* the operative indication
* the surgical procedure
* the management before and after the surgery

Patients will have a pre and post operative assessment

* Anatomical by sectional imaging
* Functional by motion analysis

Thus, it allows creating 3 digital models for the same patient:

1. Creation of Model 1: preoperative dynamic model obtained from the anatomical and functional preoperative assessment.
2. Creation of Model 2: Model 1 to which the surgery is applied according to the criteria indicated by the surgeon.
3. Creation of Model 3: a dynamic postoperative model independent of Models 1 and 2 obtained from the anatomical and functional postoperative assessment.

Validation of each model:

Each model will be compared with the patient data used to build the model, there is no comparison of patients regarding each other or models belonging to different patients. This study therefore aims to validate an individual's model on his or her own data.

* Comparison of model 1 (angle, forces, geometry) versus morphological and functional assessment before surgery
* Comparison of model 3 (angle, forces, geometry) versus morphological and functional assessment after surgery

Evaluation the surgery simulation procedure:

Comparison of model 2 (angle, forces, geometry) versus model 3

ELIGIBILITY:
Inclusion Criteria:

* If women, menopausal or on contraception if of childbearing age
* Patients who will benefit from one of the orthopedic surgical procedures corresponding to the surgeries studied
* Patient who is a member of a social security organization
* Patient who has signed a written informed consent form

Exclusion Criteria:

* Patient refusal to participate in the study
* Minor,
* Patient under guardianship and / or curators,
* Patient unable to receive information and express consent
* Pregnant and/or breastfeeding women
* Contraindication to MRI (presence of ferromagnetic materials, neurosurgical clips, vascular, pacemaker).
* Non-affiliation to a social security scheme (beneficiary or entitled person)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of simulated models regarding relative position of bones in static condition | 18 months
  comparison between real data (from imaging) vs simulated data regarding relative position of bones defining a joint:
  angles between mechanical bone axis in degree
  in two situations:
  * angles measured on pre operative imaging versus angles obtained on model 1
  * angles measured on post operative imaging versus angles obtained on model 3
Evaluation of simulated models regarding relative position of bones in dynamic condition: range of motion (ROM) | 18 months
  comparison between real data (from motion analysis) vs simulated data regarding relative position of bones defining a joint:
  total joint range of motion (ROM) projected in anatomical planes : degree of freedom of the joint (flexion, extension, abduction, adduction, medial and lateral rotation) (Kinematic parameters)
  in two situations:
  * ROM measured on pre operative motion analysis versus ROM obtained on model 1
  * ROM measured on post operative motion analysis versus ROM obtained on model 3
Evaluation of simulated models regarding forces | 18 months
  comparison between real data (from motion analysis) vs simulated data regarding kinetic parameters as forces (ground reaction forces)
  in Newton (N)
  in two situations:
  * forces measured on pre operative motion analysis versus forces obtained on model 1
  * forces measured on post operative motion analysis versus forces obtained on model 3
Evaluation of simulated models regarding moment | 18 months
  comparison between real data (from motion analysis) vs simulated data regarding kinetic parameters as joint moment
  in Newton-metre (N.m)
  in two situations:
  * moment calculated on pre operative motion analysis versus moment obtained on model 1
  * moment calculated on post operative motion analysis versus moment obtained on model 3
Evaluation of simulated models regarding pressure | 18 months
  comparison between real data (from motion analysis) vs simulated data regarding kinetic parameters as pressure (baropodometric analysis)
  in Newton per square centimeter (N/cm2)
  in two situations:
  * pressure measured on pre operative motion analysis versus pressure obtained on model 1
  * pressure measured on post operative motion analysis versus pressure obtained on model 3
comparison of post surgery changes in real and simulated results regarding bone dimension | 18 months
  comparison between real bone dimension's changes (from imaging) vs bone dimension's changes on simulated data
  difference calculated in mm
  in one situation:
  - bone dimension's difference calculated on CT scan (difference between pre and post operative bone dimensions) versus bone dimension's difference calculated on models (difference between bone dimensions obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding bone torsion | 18 months
  comparison between real bone torsion's changes (from imaging) vs bone torsion's changes on simulated data,
  difference calculated in degree
  in one situation:
  - bone torsion's difference calculated on CT scan (difference between pre and post operative bone torsions) versus bone torsion's difference calculated on models (difference between bone torsions obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding bone axis | 18 months
  comparison between real bone axis changes (from imaging) vs bone axis changes on simulated data : anatomical bone axis (corresponding mainly to the diaphyseal axis))
  difference calculated in degree
  in one situation:
  - bone axis difference calculated on imaging (difference between pre and post operative bone torsion) versus bone torsion's difference calculated on models (difference between bone torsions obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding bone volume | 18 months
  comparison between real bone volume changes (from imaging) vs bone volume changes on simulated data
  difference calculated in mm3
  in one situation:
  - bone volume difference calculated on CT scan (difference between pre and post operative bone volumes) versus bone volume difference calculated on models (difference between bone volumes obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding relative position of bones in static condition | 18 months
  comparison between real mechanical angle changes (from imaging) vs mechanical angle changes on simulated data
  difference between angles (obtained from mechanical bone axis) calculated in degree
  in one situation:
  - mechanical angle difference calculated on imaging (difference between pre and post operative mechanical angles) versus mechanical angle difference calculated on models (difference between mechanical angles obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding ROM's changes | 18 months
  comparison between real ROM'S changes (from motion analysis) vs ROM's changes on simulated data
  joint range of motion's difference calculated in degree
  in one situation:
  - ROM's difference calculated on motion analysis (difference between pre and post operative ROM) versus ROM's difference calculated on models (difference between ROM obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding moment changes | 18 months
  comparison between real moment changes (from motion analysis) vs moment changes on simulated data
  moment difference calculated in N.m
  in one situation:
  - moment difference calculated on motion analysis (difference between pre and post operative moments) versus moment difference calculated on models (difference between moments obtained on model 1 and model 3)
comparison of post surgery changes in real and simulated results regarding pressure changes | 18 months
  comparison between real pressure changes (from motion analysis) vs pressure changes on simulated data
  pressure difference calculated in N/cm2
  in one situation:
  - pressure difference calculated on motion analysis (difference between pre and post operative pressures) versus pressure difference calculated on models (difference between pressures obtained on model 1 and model 3)

SECONDARY OUTCOMES:
correlation of clinical scores and changes in function | 18 months
  changes in clinical scores (percentage) compared to the variation in the range of motion of joints studied
Comparison of post surgery models between real and simulated surgery regarding bone dimension | 18 months
  comparison between bone dimension in simulated surgery (model 2) and bone dimension in real surgery model (model 3)
  difference calculated in mm
Comparison of post surgery models between real and simulated surgery regarding bone torsion | 18 months
  comparison between bone torsion in simulated surgery (model 2) and bone torsion in real surgery model (model 3)
  difference calculated in degree
Comparison of post surgery models between real and simulated surgery regarding bone axis | 18 months
  comparison between bone axis in simulated surgery (model 2) and bone axis in real surgery model (model 3) : anatomical bone axis (corresponding mainly to the diaphyseal axis))
  difference calculated in degree
Comparison of post surgery models between real and simulated surgery regarding bone volume | 18 months
  comparison between bone volume in simulated surgery (model 2) and bone volume in real surgery model (model 3)
  difference calculated in mm3
Comparison of post surgery models between real and simulated surgery regarding point-to-surface distance of bone | 18 months
  comparison of point-to-surface distance between two pairs of bones model 1/ model 2 and model 1/model 3
  difference calculated in mm
Comparison of post surgery models between real and simulated surgery regarding relative position of bones in static condition | 18 months
  comparison between mechanical angle in simulated surgery (model 2) and mechanical angle in real surgery model (model 3)
  difference between angles (obtained from mechanical bone axis) calculated in degree
Comparison of post surgery models between real and simulated surgery regarding ROM's changes | 18 months
  comparison between ROM in simulated surgery (model 2) and ROM in real surgery model (model 3)
  joint range of motion's difference calculated in degree
Comparison of post surgery models between real and simulated surgery regarding ground reaction forces changes | 18 months
  comparison between forces in simulated surgery (model 2) and forces in real surgery model (model 3)
  ground reaction forces difference calculated in Newton
Comparison of post surgery models between real and simulated surgery regarding moment changes | 18 months
  comparison between moment in simulated surgery (model 2) and moment in real surgery model (model 3)
  moment difference calculated in N.m
Comparison of post surgery models between real and simulated surgery regarding pressure changes | 18 months
  comparison between pressure in simulated surgery (model 2) and pressure in real surgery model (model 3)
  pressure difference calculated in N/cm2
comparison of simulated joint force changes between Pre and post surgery models | 18 months
  comparison between simulated joint forces (from model 1) vs simulated joint forces (from model 2 and 3)
  joint normal contact forces difference calculated in Newton

CONTACTS AND LOCATIONS:
Overall Officials: Antoine M PERRIER, PHD, Principal Investigator — laboratoire TIMC CNRS